CLINICAL TRIAL: NCT02836938
Title: Breath Volatile Organic Compounds Patterns of Lung Transplant Patients With Chronic Lung Allograft Dysfunction
Status: Completed | Type: Observational
Sponsor: Prof. Dr. Jens Hohlfeld (Other)
Collaborators: Hannover Medical School (Other)
Responsible Party: Sponsor-Investigator, Prof. Dr. Jens Hohlfeld, Prof. Dr., Fraunhofer-Institute of Toxicology and Experimental Medicine
Organization: Fraunhofer-Institute of Toxicology and Experimental Medicine (Other)
Other Study IDs: TXVOC
Record Dates: First submitted 2016-07-05; First posted 2016-07-19 (Estimated); Last update posted 2017-02-14 (Actual); Status verified 2017-02

CONDITIONS: Chronic Lung Allograft Dysfunction (CLAD)

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (3):
- Severe: Severe chronic lung allograft dysfunction (CLAD), bronchiolitis obliterans syndrome (BOS), stage 3
  Interventions: Other: Collection of exhaled breath volatile organic compounds
- Mild: Mild chronic lung allograft dysfunction (CLAD), bronchiolitis obliterans syndrome (BOS), stage 1-2
  Interventions: Other: Collection of exhaled breath volatile organic compounds
- Control: Bronchiolitis obliterans syndrome (BOS), stage 0
  Interventions: Other: Collection of exhaled breath volatile organic compounds

INTERVENTIONS:
Other: Collection of exhaled breath volatile organic compounds

SUMMARY:
It's the aim of this study to clarify, whether the non-invasive assessment of breath can serve as a novel clinical tool to assist in the diagnosis of CLAD. If different stages of BOS can be discriminated by the level of certain VOCs than there would also be a potential to actually predict the development at an early stage and would enable an earlier intervention.

ELIGIBILITY:
Inclusion Criteria:

* Outpatient bilateral lung transplant recipients including combined transplants

Exclusion Criteria:

* Active Smoking Oxygen therapy Infection with multi or pan-resistant bacteria

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Group of transplant patients with and without signs of BOS
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2016-06; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Concentration of exhaled breath volatile organic compounds | one sample will be collected between 6 month and 20 years after lung transplantation

CONTACTS AND LOCATIONS:
Locations (1):
- Hannover Medical School, Hanover, Germany